CLINICAL TRIAL: NCT01479088
Title: Twelve-month, Multicenter, Intra-subject Controlled (Retrospective-prospective), Open-label, Active-treatment Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics (PK) of Cinacalcet Hydrochloride for the Treatment of Secondary Hyperparathyroidism (SHPT) in Paediatric Subjects With Chronic Kidney Disease (CKD) on Dialysis, Followed by 12-month Study Extension.
Brief Title: Cinacalcet in Paediatric Secondary Hyperparathyroidism (SHPT) Due to Chronic Kidney Disease (CKD)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ENRICO VERRINA (Other)
Responsible Party: Sponsor-Investigator, ENRICO VERRINA, Director of Dialysis Unit, Istituto Giannina Gaslini
Organization: Istituto Giannina Gaslini (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGG_ev_003; 2009-016797-32 (EudraCT Number)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Cinacalcet; PK; Secondary Hyperparathyroidism; Paediatric; Chronic Kidney Disease; Dialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cinacalcet tab or extemporaneous solution po added to SoC (Experimental): Subjects who meet all inclusion/exclusion criteria at baseline will be given cinacalcet 30mg film-coated tablet, for oral use added to phosphate binders and vitamin D analogue.
  For subjects receiving a cinacalcet dose <30mg, commercially available cinacalcet 30mg tab will be ground and diluted with a 5% dextrose solution. Then, an aliquot of this solution corresponding to the individually prescribed dose will be administered as indicated.
  Initial dosing of cinacalcet will be 0.5-0.75mg/kg or 30 mg po once daily (OD) each evening with food.
  During the cinacalcet dose-titration 6-month period for efficacy assessment, the dose will be increased on monthly basis by 0.5 mg/kg or by 30mg OD to achieve the target iPTH value <180 pg/mL, as tolerated by the subject, up to maximum of 180mg OD in absence of signs of hypocalcemia, according to the current summary of product characteristics.
  Interventions: Drug: Cinacalcet HCl

INTERVENTIONS:
Drug: Cinacalcet HCl — The 6-month pre-treatment period will be followed by a run-in period with a baseline evaluation prior to the drug administration, followed by a 6-month cinacalcet dose titration period, during which the dose will be increased on monthly basis by 0.5 mg/kg or by 30 mg OD up to the achievement of target iPTH value <180 pg/mL as tolerated by the patient
  Other Names: Mimpara®

SUMMARY:
Twelve-month, multicenter, intra-subject controlled (retrospective-prospective), open-label, active-treatment study to evaluate the dose-response and pharmacokinetics (PK) of cinacalcet HCl for the treatment of Secondary Hyperparathyroidism (SHPT) in paediatric subjects with chronic kidney disease (CKD) on dialysis, followed by 12-month study extension.

DETAILED DESCRIPTION:
This multicenter, intra-subject controlled, open-label, active-treatment study will assess in children affected by Secondary Hyperparathyroidism, aged 2-18 years on chronic dialysis not responsive to standard of care (SoC) therapy, the response after 6-month cinacalcet compared intra-subject to SoC alone at screening visit 6 months prior to cinacalcet start. Secondary objectives are to evaluate effects on growth over 18 months and PK profile. At baseline children have PTH levels>300 pg/mL, plasma P<6 mg/dL, and Ca 8.4-10.5 mg/dL, or Ca x P product>60 not responsive to SoC. Initial dosing of cinacalcet will be 0.5-0.75 mg/Kg per os OD to be adjusted up to a max of 180mg OD for target PTH values<180 pg/mL in absence of hypocalcemia. Thirty children will be enrolled at 12 centres participating in a national paediatric dialysis registry, corresponding to an α=0.05 and a power of 80% using the McNemar test, with an expected % of responders to cinacalcet or SoC of 40% or 5% respectively, with a drop-out rate of 15. Primary study endpoint (EP) will be the % of children who will have a reduction from baseline >25% in mean PTH levels during the 6-mo efficacy-assessment period. Among secondary EPs over 18 mos will be the % of patients with mean PTH levels<300 pg/mL; the % change in PTH, Ca, P values, and the Ca x P product; PK profile (or population profile by age) and its correlation with PTH and testosterone levels; auxological indices and growth velocity; % of children with treatment-emergent adverse events and lab abnormalities; retention on treatment and reasons of treatment withdrawal. The study will evaluate whether cinacalcet represents a safe and effective therapeutic option for SHPT children.

ELIGIBILITY:
Inclusion Criteria:

* Parents'/guardian written informed consent, and child's assent
* Age > 2 and <18 years;
* A dry body weight (BW) >10.49 Kg in males and >9.95 Kg in females, respectively;
* Inpatient or outpatient status at the time of enrolment;
* Males or females. Female subjects sexually active must be neither pregnant nor breastfeeding, and must lack childbearing potential from screening visit to the end of the safety follow-up
* On stable hemodialysis (HD) or peritoneal dialysis (PD) for their CKD for at least one month before entering the 6-month pre-treatment period;
* Plasma iPTH levels > 300 pg/mL, AND
* Plasma Ca levels > 9.4 mg/dL (with normal serum albumin level), AND
* Plasma P levels <6.5 mg/dL in patients younger than 6 years, or <6.0mg/dL in older patients, OR
* Ca x P product > 60;
* Records' availability for the following parameters 6 months prior to study entry: demographic information, physical examination, height and dry weight, auxological/anthropometric indices, blood pressure values, Kt/V urea, plasma iPTH, calcium, phosphorus, and alkaline phosphatise levels, blood pH and bicarbonate, serum creatinine/urea, C reactive protein (CRP) levels, liver function tests, blood count, blood 25(OH) vitamin D3 level.

Exclusion Criteria:

* The following laboratory values: Hb<9.0 g/dL, WBC<2000/mm3 (2x109/L), platelets <150,000/mm3 (150x109/L) only in subjects who are otherwise eligible for PK/PD assessments; abnormal liver function, defined by a total bilirubin ≥2 times the upper limit of normal values, ASAT, ALAT, γ-GT levels ≥2 times the ULN values.
* Any other lab values that in the opinion of the investigator might place the subject at unacceptable risk for participation in the study.
* History of malignancy (active malignancy, or off therapy since less than 1 year)
* History of diseases causing hypercalcemia
* Chronic inflammatory diseases (C-Reactive Protein-CRP >2 times the upper limit of normal values) requiring a concomitant corticosteroid or immunosuppressive therapy
* History of infectious diseases (including opportunistic infections) within 4 weeks prior to study entry
* Evidence as assessed by the Investigator of active or latent bacterial, viral or fungal infections at the time of potential enrollment, including subjects with evidence of HIV infection.
* Hepatitis-B surface antigen-positive subjects only in subjects who are otherwise eligible for PK/PD assessments
* Hepatitis C antibody-positive subjects who are also PCR-positive or RIBA positive only in subjects who are otherwise eligible for PK/PD assessments
* Use of recombinant human growth hormone therapy
* Use of drugs that interact with cinacalcet disposition
* Previous use of cinacalcet

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Composite EP, e.g. the proportion of patients who will have a reduction from baseline of >= 25% in mean iPTH levels with concomitant values for plasma P <6 mg/dL and Ca between 8.4 and 10.5 mg/dL or the Ca x P product <60 | 6 months
  This composite EP will address the needed information on the appropriate dose of cinacalcet to be adopted in paediatric patients, and especially in younger children, as well as on the impact of treatment with calcimimetics on serum Ca and P levels, and on SHPT control over the long term

SECONDARY OUTCOMES:
The long term control of iPTH level < 300 pg/mL | 18 months
The long term control of PTH, Ca, P, and the Ca x P product values | 18 months
The PK/ PD ( iPTH and testosterone) profile at individual patient level | 12 months
The long term auxological indices and patient growth velocity during cinacalcet treatment | 18 months
The proportion of patients with treatment-emergent adverse events (AEs), serious AEs (SAEs), and laboratory abnormalities over long term | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrico E. Verrina, MD, Principal Investigator — U.O. Nefrologia e Dialisi; Istituto di Ricovero e Cura a Carattere Scientifico Giannina Gaslini
Locations (5):
- Italy (5):
  - U.O. Nefrologia e Dialisi - Istituto di Ricovero e Cura a Carattere Scientifico Giannina Gaslini, Genoa, Italy
  - U.O. Nefrologia e Dialisi- Ospedale Giovanni XXIII, Bari
  - U.O. Nefrologia e Dialisi Pediatrica - Clinica De Marchi, Milan
  - U.O. Nefrologia e Dialisi - Ospedale Santobono, Naples
  - U.O. Nefrologia e Dialisi - Ospedale Bambino Gesù, Rome

REFERENCES:
- [Background] Klaus G, Watson A, Edefonti A, Fischbach M, Ronnholm K, Schaefer F, Simkova E, Stefanidis CJ, Strazdins V, Vande Walle J, Schroder C, Zurowska A, Ekim M; European Pediatric Dialysis Working Group (EPDWG). Prevention and treatment of renal osteodystrophy in children on chronic renal failure: European guidelines. Pediatr Nephrol. 2006 Feb;21(2):151-9. doi: 10.1007/s00467-005-2082-7. Epub 2005 Oct 25. PMID 16247644
- [Background] Silverstein DM, Kher KK, Moudgil A, Khurana M, Wilcox J, Moylan K. Cinacalcet is efficacious in pediatric dialysis patients. Pediatr Nephrol. 2008 Oct;23(10):1817-22. doi: 10.1007/s00467-007-0742-5. Epub 2008 Feb 21. PMID 18288502
- [Background] Muscheites J, Wigger M, Drueckler E, Fischer DC, Kundt G, Haffner D. Cinacalcet for secondary hyperparathyroidism in children with end-stage renal disease. Pediatr Nephrol. 2008 Oct;23(10):1823-9. doi: 10.1007/s00467-008-0810-5. Epub 2008 May 27. PMID 18504621
- [Background] Platt C, Inward C, McGraw M, Dudley J, Tizard J, Burren C, Saleem MA. Middle-term use of Cinacalcet in paediatric dialysis patients. Pediatr Nephrol. 2010 Jan;25(1):143-8. doi: 10.1007/s00467-009-1294-7. Epub 2009 Oct 17. PMID 19838738
- [Background] Harris RZ, Padhi D, Marbury TC, Noveck RJ, Salfi M, Sullivan JT. Pharmacokinetics, pharmacodynamics, and safety of cinacalcet hydrochloride in hemodialysis patients at doses up to 200 mg once daily. Am J Kidney Dis. 2004 Dec;44(6):1070-6. doi: 10.1053/j.ajkd.2004.08.029. PMID 15558528
- [Background] Padhi D, Harris RZ, Salfi M, Noveck RJ, Sullivan JT. Pharmacokinetics and pharmacodynamics of cinacalcet in hepatic impairment : phase I, open-label, parallel-group, single-dose, single-centre study. Clin Drug Investig. 2008;28(10):635-43. doi: 10.2165/00044011-200828100-00004. PMID 18783302
- [Derived] Cangemi G, Barco S, Verrina EE, Scurati S, Melioli G, Della Casa Alberighi O. Micromethod for quantification of cinacalcet in human plasma by liquid chromatography-tandem mass spectrometry using a stable isotope-labeled internal standard. Ther Drug Monit. 2013 Feb;35(1):112-7. doi: 10.1097/FTD.0b013e318278dc69. PMID 23222688
- See also: study description on the Italian Paediatric Nephrology Society website — http://www.sinp.eu/index/index/atom/131